CLINICAL TRIAL: NCT00000801
Title: Phase II Trial of Sequential Chemotherapy and Radiotherapy for AIDS-Related Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 252; ECOG E 1493
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: Vincristine; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Granulocyte Colony-Stimulating Factor; Combined Modality Therapy; Acquired Immunodeficiency Syndrome; Antineoplastic Agents, Combined; Brain Neoplasms; Lymphoma, High-Grade; Lymphoma, Intermediate-Grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Acquired Immunodeficiency Syndrome; Brain Neoplasms | interventions — Filgrastim; Vincristine; Doxorubicin; Cyclophosphamide; Cytarabine; Dexamethasone

INTERVENTIONS:
Drug: Filgrastim
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Dexamethasone

SUMMARY:
To estimate the response rate, overall and disease-free survival, toxicities, factors associated with outcome, and effect on quality of life in patients with AIDS-related primary CNS lymphoma treated with CHOD (cyclophosphamide, doxorubicin, vincristine, and dexamethasone) plus filgrastim (granulocyte-colony stimulating factor; G-CSF) and external beam irradiation. To determine other clinical markers present in this patient population.

Combined modality therapy may prove of benefit for patients with AIDS-related primary CNS lymphoma.

DETAILED DESCRIPTION:
Combined modality therapy may prove of benefit for patients with AIDS-related primary CNS lymphoma.

Patients who upon staging workup are found to be without systemic involvement undergo one cycle of chemotherapy with cyclophosphamide, doxorubicin, vincristine, dexamethasone, and G-CSF. Cyclophosphamide, doxorubicin, and vincristine are administered intravenously on day 1. Dexamethasone is administered intravenously on day 1 and then orally thereafter with gradual discontinuation. G-CSF is administered subcutaneously daily beginning on day 2 and continuing for a total of 10 days or until blood counts have recovered to an acceptable level. Patients with evidence of cancer cells in their cerebrospinal fluid (CSF) will receive chemotherapy with intrathecal cytarabine twice weekly until no further evidence of cancer cells is found in the CSF, then once weekly for 6 weeks, and then monthly for 10 months. Seven to ten days following completion of one cycle of chemotherapy, patients undergo radiotherapy to the brain at a dose of 2.5 Gy daily for 5 days per week for approximately 4 weeks. Total dose to the whole brain and meninges is 30.0 Gy in 12 fractions, and total dose to the primary boost volume is 10.0 Gy in 4 fractions. During therapy, blood is drawn weekly and brain scans are performed every 3-12 weeks. An initial CSF sample will be obtained by lumbar puncture.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Required:

* PCP prophylaxis with Bactrim, dapsone, or aerosolized pentamidine.
* Oral candidiasis prophylaxis with fluconazole, ketoconazole, or clotrimazole oral troches.
* Antiretroviral agent available by therapy IND.
* MAI prophylaxis with rifabutin (in patients with CD4 counts < 100 cells/mm3).

Patients must have:

* HIV infection.
* Primary CNS lymphoma with NO systemic involvement.

Prior Medication:

Allowed:

* Prior corticosteroids.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Concomitant malignancy other than Kaposi's sarcoma, curatively treated carcinoma in situ of the cervix, or squamous or basal cell carcinoma of the skin.
* Active uncontrolled infection.
* Renal failure, active nonmalignant duodenal ulcer, uncontrolled diabetes mellitus, or other serious medical conditions that would preclude aggressive cytotoxic chemotherapy administration.
* Active heart disease (congestive heart failure or heart block greater than first degree on EKG).

Concurrent Medication:

Excluded:

* Any investigational agent other than antiretroviral agents available by therapy IND.

Patients with the following prior conditions are excluded:

* No prior malignancy other than Kaposi's sarcoma, curatively treated carcinoma in situ of the cervix, or squamous cell or basal cell carcinoma of the skin.
* No new infectious complications within the past 2 weeks that require a change in antibiotics.
* History of myocardial infarction within the past 3 months.

Prior Medication:

Excluded:

* Prior chemotherapy other than for Kaposi's sarcoma.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krigel RL, Study Chair; Von Roenn J, Study Chair
Locations (7):
- United States (7):
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - ECOG Data Management Office, Brookline, Massachusetts
  - Mount Sinai Med Ctr, New York, New York
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Schultz C, Scott C, Sherman W, Donahue B, Fields J, Murray K, Fisher B, Abrams R, Meis-Kindblom J. Preirradiation chemotherapy with cyclophosphamide, doxorubicin, vincristine, and dexamethasone for primary CNS lymphomas: initial report of radiation therapy oncology group protocol 88-06. J Clin Oncol. 1996 Feb;14(2):556-64. doi: 10.1200/JCO.1996.14.2.556. PMID 8636771